CLINICAL TRIAL: NCT04609878
Title: A Randomized, Double-Blind, Double Dummy, Parallel Group, Multicenter Variable Length Study to Assess the Efficacy and Safety of PT010 Relative to PT009 and Symbicort® in Adult and Adolescent Participants With Inadequately Controlled Asthma
Brief Title: Study to Assess PT010 in Adult and Adolescent Participants With Inadequately Controlled Asthma (KALOS)
Acronym: KALOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5982C00007; 2023-505787-11 (Registry Identifier: CTIS); 2020-001520-34 (EudraCT Number)
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Budesonide, glycopyrronium, and formoterol fumarate (BGF) MDI 320/28.8/9.6 μg (Experimental): BGF MDI 320/28.8/9.6 μg Budesonide, glycopyrronium, and formoterol fumarate (PT010) Metered Dose Inhaler (MDI)
  Interventions: Drug: BGF MDI 320/28.8/9.6 μg
- BGF MDI 320/14.4/9.6 μg (Experimental): BGF MDI 320/14.4/9.6 μg Budesonide, glycopyrronium, and formoterol fumarate (PT010) Metered Dose Inhaler (MDI)
  Interventions: Drug: BGF MDI 320/14.4/9.6 μg
- Budesonide and formoterol fumarate (BFF) MDI 320/9.6 μg (Active Comparator): BFF MDI 320/9.6 μg (Experimental/Comparator) Budesonide and formoterol fumarate (PT009) Metered Dose Inhaler (MDI)
  Interventions: Drug: BFF MDI 320/9.6 μg
- Symbicort® (Active Comparator): Budesonide/ formoterol fumarate pressurized metered dose inhaler (pMDI) 320/9 μg
  Interventions: Drug: BFF pMDI 320/9 μg

INTERVENTIONS:
Drug: BGF MDI 320/28.8/9.6 μg — Budesonide, glycopyrronium, and formoterol fumarate metered dose inhaler
  Other Names: BGF
  Arms: Budesonide, glycopyrronium, and formoterol fumarate (BGF) MDI 320/28.8/9.6 μg
Drug: BGF MDI 320/14.4/9.6 μg — Budesonide, glycopyrronium, and formoterol fumarate metered dose inhaler
  Other Names: BGF
  Arms: BGF MDI 320/14.4/9.6 μg
Drug: BFF MDI 320/9.6 μg — Budesonide and formoterol fumarate metered dose inhaler
  Other Names: BFF
  Arms: Budesonide and formoterol fumarate (BFF) MDI 320/9.6 μg
Drug: BFF pMDI 320/9 μg — Budesonide/formoterol fumarate pressurized metered dose inhaler
  Other Names: Symbicort®
  Arms: Symbicort®

SUMMARY:
This is a variable length study to evaluate the efficacy and safety of budesonide/glycopyrronium/formoterol inhaler in adults and adolescents with severe asthma inadequately controlled with standard of care

DETAILED DESCRIPTION:
This is a randomized, double-blind, double dummy, parallel group, multicenter 24 to 52 week variable length study to assess the efficacy and safety of budesonide, glycopyrronium, and formoterol fumarate metered dose inhaler (MDI) relative to budesonide and formoterol fumarate MDI and Symbicort® pressurized MDI in adult and adolescent participants with inadequately controlled asthma. Approximately 2200 participants will be randomized globally.

ELIGIBILITY:
Inclusion Criteria:

1. 12 to 80 years of age, male and female, BMI <40 kg/m2; females must be not of childbearing potential or using a form of highly effective birth control.
2. Documented history of physician-diagnosed asthma > and/or = 1 year prior to V1.
3. Regularly using a stable daily ICS/LABA regimen (including a stable ICS dose) with medium-to-high ICS doses for at least 4 weeks prior to V1.
4. ACQ-7 total score ≥1.5 at Visits 1, 3, and 5 (pre-randomization).
5. FEV1 % (assessed as an average of the 60 and 30 minute pre-dose assessments) predicted normal at V1, 2, 3, 4, and 5 (pre-randomization)

   * Participants ≥ 18 years of age: < 80%
   * Participants 12 to <18 years of age: < 90%
6. FEV1 post-albuterol at V2 or V3 (if repeat needed).

   * Participants > and/or = 18 years of age: Increase > and/or = 12% and > and/or = 200 mL.
   * Participants 12 to <18 years of age: Increase =12% either in the 12 months prior to Visit 1 or at Visit 2, or at Visit 3.
   * Note: Even if there is documented history of reversibility, all participants must be assessed for reversibility at Visit 2 (and Visit 3, if reversibility is not demonstrated at Visit 2) to provide reversibility baseline data for characterization.
7. Willing and, in the opinion of the Investigator, able to adjust current asthma therapy, as required by the protocol.
8. Demonstrate acceptable MDI/pMDI administration technique.
9. Received no asthma medication other than run-in BFF MDI BID and albuterol as needed during screening (except for allowed medications as defined in Table 9 and systemic corticosteroid or ICS for the treatment of an asthma exacerbation).
10. eDiary 14-day compliance ≥70% during screening (defined as completing the daily eDiary for any 10 mornings and any 10 evenings and answering "Yes" to taking 2 puffs of run-in BFF MDI for any 10 mornings and 10 evenings in the last 14 days prior to randomization).
11. No respiratory infection in the 4 weeks prior to randomization, or asthma exacerbation treated with systemic corticosteroid and/or additional ICS treatment in the 4 weeks prior to randomization.

Exclusion Criteria:

1. Completed treatment for respiratory infection or asthma exacerbation with systemic corticosteroids within 4 weeks of V1.

2a. Participants where, in the opinion of the Investigator, treatment with biological therapy for asthma would be appropriate.

2b. Any marketed or investigational biologics within 3 months or 5 half-lives of V1, whichever is longer and must not be used during study duration.

3. Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months prior to V1 (including all forms of tobacco, e-cigarettes or other vaping devices, and marijuana).

4. Current evidence of Chronic Obstructive Pulmonary Disease (COPD).

5a. Oral and IV corticosteroid use (any dose) within 4 weeks of V1.

5b. Use of systemic corticosteroids for any other reason except for the acute treatment of severe asthma exacerbation is prohibited for the duration of the study.

5c. Depot corticosteroid use for any reason within 3 months of V1.

6. Use of Long-Acting Muscarinic Antagonist (LAMA), either alone or as part of an inhaled combination therapy, in the 12 weeks prior to V1.

7. Use of oral beta2-agonist within 3 months of V1.

8. Use of any immunomodulators or immunosuppressive medication within 3 months or 5 half-lives, whichever is longer, and must not be used during the study duration.

9. Narrow angle glaucoma not adequately treated and/or change in vision that may be relevant, in the opinion of the Investigator, within 3 months of Visit 1.

10. Life-threatening asthma defined as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s).

11. Hospitalization for asthma within 2 months of Visit 1.

12. Known history of drug or alcohol abuse within 12 months of Visit 1.

13. Regular use of a nebulizer or a home nebulizer for receiving asthma medications.

14. Using any herbal products by inhalation or nebulizer within 4 weeks of Visit 1 and does not agree to stop during the study duration.

15. Participation in another clinical study with a study intervention administered in the last 30 days or 5 half-lives, whichever is longer. Any other study intervention that is not identified in the protocol is prohibited for use during study duration.

16. Participants with a known hypersensitivity to beta2-agonists, corticosteroids, anticholinergics, or any component of the MDI or pMDI.

17. Study Investigators, sub-Investigators, coordinators, and their employees or immediate family members.

18. For women only - currently pregnant (confirmed with positive highly sensitive pregnancy test), breast-feeding, or planned pregnancy during the study or not using acceptable contraception measures, as judged by the Investigator.

Please refer to the study protocol for the complete inclusion and exclusion criteria list.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2274 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in forced expiratory volume in 1 second (FEV1) area under the curve 0 to 3 hours (AUC0-3) at Week 24 | 24 Weeks
  Change from baseline in forced expiratory volume in 1 second (FEV1) area under the curve 0 to 3 hours (AUC0-3) at Week 24
Rate of severe asthma exacerbations | Up to 52 weeks
  Primary end point(s) of Pooled Studies D5982C00007 and D5982C00008: Rate of severe asthma exacerbations

SECONDARY OUTCOMES:
Change from baseline in morning pre-dose trough FEV1 at Week 24 | 24 Weeks
  Change from baseline in morning pre-dose trough FEV1 at Week 24
Percentage of responders in Asthma Control Questionnaire (ACQ)-7 (≥0.5 decrease equals response) at Week 24 | 24 weeks
  Percentage of responders in ACQ-7 (≥0.5 decrease equals response) at Week 24. Additional analysis will be conducted using pooled data from studies D5982C00007 and D5982C00008
Percentage of responders in ACQ-5 (≥0.5 decrease equals response) at Week 24 | 24 Weeks
  Percentage of responders in ACQ-5 (≥0.5 decrease equals response) at Week 24. Additional analysis will be conducted using pooled data from studies D5982C00007 and D5982C00008
Percentage of responders in the Asthma Quality of Life Questionnaire for 12 years and older (AQLQ +12) (≥0.5 increase equals response) at Week 24 | 24 weeks
  Percentage of responders in the Asthma Quality of Life Questionnaire for 12 years and older (AQLQ(s) +12) (≥0.5 increase equals response) at Week 24. Additional analysis will be conducted using pooled data from studies D5982C00007 and D5982C00008
Percentage of responders in the St. George's Respiratory Questionnaire (SGRQ) (≥4.0 unit decrease equals response) at Week 24 | 24 Weeks
  Percentage of responders in the St. George's Respiratory Questionnaire (SGRQ) (≥4.0 unit decrease equals response) at Week 24
Onset of action on Day 1: Absolute change in FEV1 at 5 minutes on Day 1 | Day 1
  Onset of action on Day 1: Absolute change in FEV1 at 5 minutes on Day 1
Time to first severe asthma exacerbation | Up to 52 Weeks
  Secondary end point(s) of Pooled Studies D5982C00007 and D5982C00008:
  Time to first severe asthma exacerbation
Rate of moderate/severe asthma exacerbations | Up to 52 Weeks
  Secondary end point(s) of Pooled Studies D5982C00007 and D5982C00008:
  Rate of moderate/severe asthma exacerbations
Time to first moderate/severe asthma exacerbation | Up to 52 Weeks
  Secondary end point(s) of Pooled Studies D5982C00007 and D5982C00008:
  Time to first moderate/severe asthma exacerbation
Rate of severe asthma exacerbations for participants with percent predicted FEV1 ≤ 55% at baseline. | Up to 52 Weeks
  Secondary end point(s) of Pooled Studies D5982C00007 and D5982C00008: Rate of severe asthma exacerbations for participants with percent predicted FEV1 ≤ 55% at baseline.
Rate of severe asthma exacerbations for participants with ≥ 1 severe exacerbation in the 12 months prior to Visit 1. | Up to 52 Weeks
  Secondary end point(s) of Pooled Studies D5982C00007 and D5982C00008: Rate of severe asthma exacerbations for participants with ≥ 1 severe exacerbation in the 12 months prior to Visit 1.

CONTACTS AND LOCATIONS:
Locations (287):
- United States (99):
  - Research Site, Saraland, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Sun City West, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Covina, California
  - Research Site, Encinitas, California
  - Research Site, Fresno, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Hills, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Thousand Oaks, California
  - Research Site, Upland, California
  - Research Site, Westminster, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, Brandon, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Adairsville, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Tyrone, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, River Forest, Illinois
  - Research Site, Brownsburg, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Crowley, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Potomac, Maryland
  - Research Site, Waldorf, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Hannibal, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Toms River, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New Hyde Park, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Denver, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Grants Pass, Oregon
  - Research Site, DuBois, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Boerne, Texas
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Harlingen, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Nederland, Texas
  - Research Site, Pearland, Texas
  - Research Site, Red Oak, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Spring, Texas
  - Research Site, Tomball, Texas
  - Research Site, Ogden, Utah
  - Research Site, West Valley City, Utah
  - Research Site, Colchester, Vermont
  - Research Site, Manassas, Virginia
  - Research Site, Kingwood, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Cudahy, Wisconsin
- Argentina (10):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Fernando
- Belgium (2):
  - Research Site, Liège
  - Research Site, Namur
- Bulgaria (17):
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Kozloduy
  - Research Site, Lovech
  - Research Site, Pazardzhik
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vidin
  - Research Site, Vratsa
- Canada (13):
  - Research Site, Edmonton, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- Chile (4):
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
- Hungary (10):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Encs
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Komárom
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szigetvár
- India (12):
  - Research Site, Ahmedabad
  - Research Site, Aligarh
  - Research Site, Belagavi
  - Research Site, Coimbatore
  - Research Site, Dehradun
  - Research Site, Gūrgaon
  - Research Site, Jaipur
  - Research Site, Mohali
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Thane
  - Research Site, Visakhapatnam
- Italy (7):
  - Research Site, Bari
  - Research Site, Casatenovo
  - Research Site, Cona
  - Research Site, Monserrato
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
- Japan (39):
  - Research Site, Chino-shi
  - Research Site, Chūōku
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Habikino-shi
  - Research Site, Hamamatsu
  - Research Site, Higashiibaraki-gun
  - Research Site, Himeji-shi
  - Research Site, Hiroshima-shi, Naka-ku
  - Research Site, Hitachi-Naka
  - Research Site, Ikoma-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kitakyushu
  - Research Site, Kiyose-shi
  - Research Site, Kokubunji-shi
  - Research Site, Kyoto
  - Research Site, Meguro-ku
  - Research Site, Nagoya
  - Research Site, Nankoku-shi
  - Research Site, Obihiro
  - Research Site, Omuta-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Sakaide-shi
  - Research Site, Sapporo
  - Research Site, Setagaya-ku
  - Research Site, Shibuya-ku
  - Research Site, Shimotsuga-gun
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takarazuka-shi
  - Research Site, Tanabe-shi
  - Research Site, Toon-shi
  - Research Site, Toshima-ku
  - Research Site, Tsuchiura-shi
  - Research Site, Utsunomiya
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- New Zealand (6):
  - Research Site, Auckland
  - Research Site, Grafton
  - Research Site, Nawton
  - Research Site, Nelson
  - Research Site, Rotorua
  - Research Site, Wellington
- Peru (2):
  - Research Site, Lima
  - Research Site, Piura
- Philippines (9):
  - Research Site, Baguio City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Lipa City
  - Research Site, Los Baños
  - Research Site, Manila
  - Research Site, Marilao
  - Research Site, Quezon City
- Poland (15):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Częstochowa
  - Research Site, Karczew
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Piaseczno
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Sosnowiec
  - Research Site, Strzelce Opolskie
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Wroclaw
- Puerto Rico (3):
  - Research Site, Caguas
  - Research Site, Guaynabo
  - Research Site, San Juan
- Romania (3):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Timișoara
- South Korea (7):
  - Research Site, Cheongju-si
  - Research Site, Gangwon-do
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
  - Research Site, Ulsan
- Spain (11):
  - Research Site, Barcelona
  - Research Site, Benalmádena
  - Research Site, Coslada
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Málaga
  - Research Site, Pozuelo de Alarcón
  - Research Site, Santander
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (7):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (7):
  - Research Site, Bang Kra So
  - Research Site, Bangkok
  - Research Site, Chanthaburi
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Mueang
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162